CLINICAL TRIAL: NCT02226107
Title: Training Latinos as Peer Patient Navigators for Colon Cancer Screening
Brief Title: Latino Peers as Patient Navigators for Colon Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 11-1374
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Colon Cancer
Keywords: Lay health worker; Patient navigation; Screening colonoscopy; Colon cancer; Training; Hispanic; Latino
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer-PN (Experimental): Peer Patient Navigation
  Interventions: Behavioral: Peer-PN
- Pro-PN (Active Comparator): Professional Patient Navigation
  Interventions: Behavioral: Pro-PN

INTERVENTIONS:
Behavioral: Peer-PN — Participants in the peer-PN group will also receive two navigation telephone calls: 1) to schedule the colonoscopy, and 2) a reminder call one week before the procedure. It is expected that these phone calls will be shortly longer than the Pro-PN calls by 5-7 minutes because of the additional focus on culture and peer modeling. Peers will remind the patient about the procedure and address concerns, but will provide culturally specific, identity-based navigation, in which they will speak specifically about Latino rates of CRC screening while also modeling self-efficacy by describing what their experience was like before, during and after the colonoscopy procedure.
  Other Names: Peer Patient Navigation
  Arms: Peer-PN
Behavioral: Pro-PN — Participants in the standard navigation group receive two phone calls: 1) to schedule the colonoscopy and 2) a reminder call one week before the procedure. The phone calls will each last approximately 15 minutes. During the second phone call, the patient will be reminded about the procedure and any concerns they may have will be addressed. Professional navigators will also be advised to not disclose their race or ethnicity or to discuss specific issues related to Latinos and CRC screening.
  Other Names: Professional Patient Navigation
  Arms: Pro-PN

SUMMARY:
Disparities among racial and ethnic minorities remain prevalent despite advances in medical science that make thes early detection and prevention of colorectal cancer a possibility for all human kind. It is estimated that 90% of colorectal cancer deaths could be prevented through screening. Unfortunately, among Latinos, colorectal cancer is the second leading cause of cancer death. This rate is influenced by the fact that Latinos have the lowest rates of colorectal cancer screening compared to other US racial groups. Moreover, Latinos are more likely than whites to be diagnosed with advanced-stage colorectal cancer, when treatment options are more limited. Lay health worker interventions for breast and cervical cancer education and screening have demonstrated success in increasing both knowledge and screening rates among racial and ethnic minorities. Additionally, our research has also shown success in training African Americans as peer navigators to increase colorectal cancer screening. Few lay health interventions, however, have been designed specifically for colorectal cancer screening among Latinos. Thus, the purpose of this study is to expand peer navigation for colorectal cancer screening to Latinos and increase their participation in screening by training Latinos, who have had a colonoscopy, to help navigate other Latinos through the colonoscopy screening procedure.

This study will focus on expanding the work of our research group by training Latino peers, who are 50 years or older, have had a colonoscopy, and can model successful colonoscopy screening completion to navigate Latino patients for screening. First, a training manual will be developed which will be culturally specific to Latinos. Feedback and input from community members will guide the development of the manual and training program. Second, the training program will be carried out with six bilingual Latino peers, who will be taught to master the core skills of patient navigation for screening colonoscopy. Finally, we will gather preliminary information about the trained peers' ability to successfully navigate patients for colonoscopy screening. If successful, this training program has the potential to increase colonoscopy screening rates of Latinos and will be critical to the development of future large-scale in interventions aimed at reducing advanced stage diagnosis of colorectal cancer and ultimately colorectal cancer deaths among Latinos.

DETAILED DESCRIPTION:
Patients are being referred and scheduled for screening and diagnostic colonoscopy as part of standard of care.

For research purposes, participants will be randomized to one of two kinds of patient navigation:

1. Standard patient navigation (Pro-PN) receiving care that they would normally receive if they were not participating in the study with patient navigation from the primary mentor's staff.
2. Peer Patient Navigation (Peer-PN): Participants will be assisted by Latino/Hispanic peers who have undergone colonoscopy, and are able to discuss, first-hand, their personal experience undergoing colonoscopy and describe how they coped effectively with the procedure. Medical advice will not be given.

Both groups will receive 3 intervention phone calls from their assigned navigators: 1) to schedule the colonoscopy 2) a reminder call two weeks before the procedure and 3) a reminder call three days before the procedure. PPN's will undergo three months of training supervised by Dr. Sly (who will be mentored/supervised by Dr. Itzkowitz and Professor Jandorf). Multiple modes of training will be used (didactic discussion, observation, role-playing, one-on-one sessions, ongoing feedback, rehearsal, supervision (by study investigator and mentors) via review of audio-tape recordings of Latino peers' navigation phone calls to the participants and a take-home training manual).

Patients receiving standard patient navigation will receive the care and assessments that they would normally receive if they were not participating in a study. Patients in the Peer-PN group will be guided through the colonoscopy process by a Latino/Hispanic peer who has undergone colonoscopy and will provide the personal prospective of how they coped with the procedure.

At some point before the colonoscopy procedure, patients will receive a phone call, during which a research assistant will administer a questionnaire in the form of an interview. Study staff will assess health care behavior, fear of colonoscopy and concerns about CRC screening, medical mistrust, interpersonal communication, social influence, and self-efficacy. A medical chart review will also be completed after the colonoscopy for all patients to assess completion of the examination as well as prep quality and any findings where additional clinical follow-up was required. Colonoscopy results will also be collected to assess quality of care and measure the efficacy of Peer-PN navigations compared to standard navigation, particularly potential differences based on study group, i.e., compliance. No other information outside of standard of care will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a screening or diagnostic colonoscopy by a primary care physician
* 50 years or older
* Identify as Hispanic or Latino
* Provide informed consent in Spanish or English
* Have access to a working telephone

Exclusion Criteria:

* Personal history of colon cancer
* Personal history of any chronic gastrointestinal disorder (i.e., colitis, irritable bowel syndrome)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Colonoscopy Completion | up to 4 months
  Participants will be given up to four months (including re-scheduling) to complete their colonoscopy after an initial appointment is scheduled.

CONTACTS AND LOCATIONS:
Overall Officials: Jamilia Sly, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States